CLINICAL TRIAL: NCT02608580
Title: Survey in a Population of Sickle Cell Disease Patients to Evaluate the Transition Between the Queen Fabiola Children Hospital and the CHU Brugmann Hospital, and the Quality of the Hospital Care Within the CHU Brugmann Hospital.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Andre Efira, Head of Clinic, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUB-Transition
Record Dates: First submitted 2015-11-17; First posted 2015-11-18 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Sickle Cell Disease
Keywords: pediatric hospital care; adult hospital care; sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with sicke cell disease (Other): Adult sickle cell disease patients will fill in a survey about the quality of their hospital care, in the transition period between the pediatric to an adult hospital care system.
  Since filling in this survey is not part of the standard of care, this study has been defined as interventional.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey

SUMMARY:
Sickle cell disease is a genetic disease responsible for an abnormal hemoglobin.The anomaly has several consequences: a low hemoglobin rate (chronic anemia), plugs formed by red blood cells in blood vessels (extremely painful vaso-occlusive crises) and greater susceptibility to infections.

Patients with this disease should be monitored medically continuously from birth. At adulthood, they will pass from a pediatric medical care system to an adult medical care system.This transition can be experienced with more or less ease, depending on the organization within the pediatric and adult hospitals.

This questionnaire aims to assess the quality of the transition between pediatric and adult services.The investigators want to better estimate hospital work and improve the quality of care for this type of patients, throughout their entire medical history.

DETAILED DESCRIPTION:
Sickle cell disease is a genetic disease responsible for an abnormal hemoglobin. It particularly affects populations with an African ascent (300 000 African children are born every year with this genetic anomaly).

The anomaly has several consequences: a low hemoglobin rate (chronic anemia), plugs formed by red blood cells in blood vessels (extremely painful vaso-occlusive crises) and greater susceptibility to infections.

The severity of sickle cell disease is variable among children. Some develop frequent and serious complications, while others don't. A child with sickle cell disease is hospitalized about a week a year in average (for a painful crisis, infection or worsening of anemia).

Patients with this disease should be monitored medically continuously from birth. At adulthood, they will pass from a pediatric medical care system to an adult medical care system.This transition can be experienced with more or less ease, depending on the organization within the pediatric and adult hospitals.

This questionnaire aims to assess the quality of the transition between pediatric and adult services.The investigators want to better estimate hospital work and improve the quality of care for this type of patients throughout their entire medical history.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease patients, beeing admitted in the CHU Brugmann Hospital (Horta site) after having been followed in the Queen Fabiola Children Hospital.

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Factors impacting the quality of transition between the pediatric and adult care system | 1 day at the first scheduled hospital visit within the CHU Brugmann (according to standard of care for adults)
  The factors will be evaluated with a survey (questionnaire to be filled in)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Agnès Azerad, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium